CLINICAL TRIAL: NCT01425229
Title: Influence of OATP1B1 and CYP2C9 Genotypes on the Pharmacokinetics of Steady State Bosentan Before and During CYP3A4-inhibition by Clarithromycin
Brief Title: Influence of OATP1B1 and CYP2C9 Genotypes on the Pharmacokinetics of Bosentan Before and During Clarithromycin
Status: Completed | Type: Observational
Sponsor: Gerd Mikus (Other)
Responsible Party: Sponsor-Investigator, Gerd Mikus, Prof. Dr. med. Gerd Mikus, Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: K318; 2010-021392-93 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Drug Interactions
Keywords: steady state; bosentan; clarithromycin
MeSH Terms: interventions — Bosentan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bosentan: Haplotypes of CYP2C9 and OATP1B1 characterisation of CYP2C9 (CYP2C9*2 (rs1799853), CYP2C9*3 (rs1057910)) and OATP1B1 (SLCO1B1*15 (rs2306283, rs4149056))
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — * Administration of bosentan: 1 x 125 mg p.o. on day 1, 2 x 125 mg p.o. on day 2-14
  * Administration of clarithromycin: 2 x 500 mg p.o. on day 11-14
  Other Names: Tracleer

SUMMARY:
The aim of the present study is to assess the impact of the OATP1B1 genotype (SLCO1B1*15 vs. wild type; ~2% SLCO1B1*15 haplotypes in Caucasian population) and the CYP2C9 genotype (*2 and *3 allele vs. wild type; ~5% poor metabolisers in Caucasian population) on the pharmacokinetics of bosentan and the impact of CYP3A4-inhibition by clarithromycin on steady state bosentan which is a CYP3A4 inducer itself.

This study will focus on differential effects of genotypes and co-medication on the pharmacokinetics of bosentan at the metabolic and transport level. Participants will be genotyped for CYP2C9 (inclusion criterion), OATP1B1 (inclusion criterion), and CYP3A5 (no inclusion criterion).

ELIGIBILITY:
Inclusion Criteria:

* Good state of health (physically and mentally)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Voluntarily signed informed consent after full explanation of the study to the participant.
* No clinically relevant findings in any of the investigations of the pre-study examination, especially aminotransferase elevations ≥ 3 × ULN. Minor deviations of other laboratory values from normal range may be acceptable, if judged by the investigator to be of no clinical relevance.
* Known genotype for CYP2C9 and OATP1B1 polymorphism.
* Agreement to abstain from alcoholic beverages during the time of the study.
* Females must agree to use a reliable contraception (Pearl Index <1%), e.g. double barrier method.

Exclusion Criteria:

* Any regular drug treatment within the last two months, except for oral contraceptives in female volunteers and L-thyroxine.
* Any intake of a substance known to induce or inhibit drug metabolising enzymes or drug transporters within a period of less than 10 times the respective elimination half-life or 2 weeks, whatever is longer
* Any participation in a clinical trial within the last month before inclusion
* Any physical disorder which could interfere with the participant's safety during the clinical trial or with the study objectives
* Any acute or chronic illness, or clinically relevant findings in the pre-study examination, especially: a) any condition, which could modify absorption, distribution, metabolism, or excretion of the drug regimen under investigation b) Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Regular smoking
* Blood donation within 6 weeks before first study day
* Excessive alcohol drinking (more than approximately 20 g alcohol per day)
* Inability to communicate well with the investigator due to language problems or poor mental development
* Inability or unwillingness to give written informed consent
* Known or planned pregnancy or breast feeding
* Pre-existing moderate or severe liver impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, Prof. Dr., Principal Investigator — deputy head of department
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Dingemanse J, van Giersbergen PL. Clinical pharmacology of bosentan, a dual endothelin receptor antagonist. Clin Pharmacokinet. 2004;43(15):1089-115. doi: 10.2165/00003088-200443150-00003. PMID 15568889

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosentan: Bosentan pharmacokinetics
Period: Bosentan Single Dose
Arm/Group | Bosentan
Started | 16
Completed | 16
Not Completed | 0
Period: Bosentan Steady-state
Arm/Group | Bosentan
Started | 16
Completed | 16
Not Completed | 0
Period: Bosentan During Clarithromycin
Arm/Group | Bosentan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bosentan: Bosentan PK
Arm/Group | Bosentan
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  Germany | 16

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: AUC of bosentan after first-dose, at steady-state and during clarithromycin therapy
Time Frame: 0-infinity; dosing interval
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/ml
Groups:
- Bosentan After First Dose: administration of bosentan 125 mg p.o. single dose
- Bosentan at Steady-state: administration of bosentan 125 mg p.o. b.i.d. on day 2-10
- Bosentan During Clarithromycin: administration of bosentan 125 mg p.o. b.i.d. on day 11-14 and administration of clarithromycin 500 mg p.o b.i.d. on day 11-14
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During Clarithromycin
Number analyzed (Participants) | 16 | 16 | 16
h*ng/ml | 11900 [9730 to 14500] | 6830 [5330 to 8750] | 25500 [21700 to 29900]

2. Primary Outcome: Cmax
Description: Cmax after the first dose of bosentan, at steady-state, during clarithromycin
Time Frame: after first dose, at steady-state, during clarithromycin
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During Clarithromycin
Number analyzed (Participants) | 16 | 16 | 16
ng/ml | 1890 [1540 to 2310] | 1460 [1120 to 1900] | 5570 [4600 to 6740]

ADVERSE EVENTS:
Groups:
- Bosentan After First Dose: Bosentan PK after first dose
- Bosentan at Steady-state: Bosentan PK at steady-state
- Bosentan During Clarithromycin: Bosentan PK during clarithromycin
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 9/16 | 9/16 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan After First Dose (N=16) | Bosentan at Steady-state (N=16) | Bosentan During Clarithromycin (N=16)
Xerostomia (Gastrointestinal disorders) | 0 | 0 | 1
Nasopharyngitis (General disorders) | 3 | 3 | 2
Nasal congestion (General disorders) | 4 | 4 | 1
Headache (General disorders) | 5 | 4 | 5
Loss of apetite (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Night sweats (General disorders) | 1 | 1 | 0
Dizziness (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 1 | 1 | 1
Epigastric pain (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
increase of creatinine kinase (Investigations) | 0 | 0 | 1
Increase of aspartate transaminase (Investigations) | 0 | 0 | 1
taste disorder (General disorders) | 0 | 0 | 1
concentration difficulty (General disorders) | 0 | 0 | 1
Tachykardia (Investigations) | 0 | 0 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
tinnitus (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No